CLINICAL TRIAL: NCT04497974
Title: Role of Long-term Dietary Sweetness Exposure on Sweetness Preferences
Brief Title: Sweet Tooth: Nature or Nurture? Role of Long-term Dietary Sweetness Exposure on Sweetness Preferences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Bournemouth University (Other); TKI Agri & Food (Unknown); Next Food Collective (Unknown); American Beverage Association (Other); Arla Foods (Industry); Cargill (Industry); Firmenich, Switzerland (Unknown); International Sweeteners Association (Unknown); SinoSweet, China (Unknown); Cosun Nutrition Center, Netherlands (Unknown); Unilever R&D (Industry)
Responsible Party: Principal Investigator, Monica Mars, Associate Professor dr.ir Monica Mars, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL72134.081.19
Record Dates: First submitted 2019-12-16; First posted 2020-08-04 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Food Preferences
Keywords: sweetness; preferences
MeSH Terms: conditions — Food Preferences | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Randomised controlled intervention study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular dietary sweetness exposure - Control (Active Comparator): Regular dietary sweetness exposure (RSE) - The RSE group consumes a diet with 25 - 30 % energy from sweet tasting foods, for 6 months.
  Interventions: Other: Dietary intervention
- Low dietary sweetness exposure - Experimental (Experimental): Low dietary sweetness exposure (LSE) - The LSE group consumes a diet with 10 - 15 % energy from sweet tasting foods, for 6 months.
  Interventions: Other: Dietary intervention
- High dietary sweetness exposure - Experimental (Experimental): High dietary sweetness exposure (HSE) - The HSE group consumes a diet with 40 - 45 % energy from sweet tasting foods, for 6 months.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Varying the exposure to sweetness via diet manipulation.

SUMMARY:
In recent years, social pressure has been exerted towards lowering sugar and sweetness levels in foods, with the aim of decreasing the sweetness preference of the general population. However, the resilience/flexibility of sweetness preferences and the impact on energy intake is a fundamental knowledge gap. Recent, relatively long-term studies limited to no more than 3 months did not find a relationship between sweetness exposure and sweetness preferences. Therefore, a longer-term systematic investigation is necessary to objectively evaluate whether sweetness preferences can be altered via varying the sweetness exposure and whether it can affect other outcomes, such as perceived taste intensity, food intake, body weight, body composition, glucose homeostasis and sweet liker type. The study sample will consist of 180 subjects. Enrolled participants will be distributed into three intervention groups; regular dietary sweetness exposure (n=60); low dietary sweetness exposure (n=60); and high dietary sweetness exposure (n =60). The intervention is semi-controlled for a period of six months. Preference and perceived taste intensity of a series of familiar and unfamiliar foods will be assessed at baseline (Day 0), during the intervention (Month 1, Month 3, Month 6) and in the follow-up period (Month 7, Month 10). Furthermore, outcomes such as observed food choice and intake during a test meal, reported food preferences, reported food cravings, sweet-liker type, glucose homeostasis, body weight, body composition and biomarkers related to diabetes and cardiovascular disease will be assessed as well.

DETAILED DESCRIPTION:
Evidence supporting sweetness preference alterations via variations in dietary sweetness exposure is limited. Most studies investigating this focused only on specific sweet elements in the diet, (e.g. beverages; mono- and disaccharides; high-energy dense snacks) instead of sweetness in the diet as a whole. Furthermore, there is no clear evidence about the relation between dietary sweetness exposure and weight gain. Therefore, longer term, sufficiently-powered studies with a 'whole diet' approach are needed to address the question whether sweet preferences can be altered (suppressed or stimulated) by variations in sweetness exposure. It is important to answer this question so that dietary recommendations can be scientifically tailored accordingly. The present study will provide breakthrough evidence about the flexibility/adaptability of sweetness preferences, in terms of effect sizes and direction, duration of effects, and impact on dietary intake, glucose homeostasis and body weight. This information is particularly relevant for product development by food industries in the context of reformulation strategies, and for governments to base their dietary guidelines upon.

The primary study objective is to assess the effect of a 6-month low, regular and high dietary sweetness exposure on sweetness preference in a series of familiar and unfamiliar foods. Preference will be assessed in both familiar and unfamiliar foods since, preferences in familiar, commonly eaten foods might by harder to change compared to those for unfamiliar foods, because there is no consumer-expected sweetness level associated with unfamiliar foods. The secondary objective is to assess the effect of a 6-month low, regular and high dietary sweetness exposure on sweetness perception, food choice and intake during a test meal, dietary taste patterns, taste preferences, food cravings, sweet-liker type, glucose homeostasis, biomarkers related to cardiovascular disease (CVD) and diabetes, body weight and body composition. Participants will be matched on age, gender, BMI and sweet liker status and randomly allocated to one of the three intervention arms: (1) regular dietary sweetness exposure (25-30 percent daily energy from sweet foods) (control) (n=60); (2) low dietary sweetness exposure (10-15 percent daily energy from sweet foods) (n=60); and (3) high dietary sweetness exposure (40-45 percent daily energy from sweet foods) (n=60). The intervention is semi-controlled, meaning that 50 percent of the foods will be provided to participants. Foods are offered ad libitum, on a weekly basis and macronutrient composition of the offered foods is similar in energy and macronutrient composition, that is fat, protein, carbohydrates and fibres, but different in sweetness. New methodology of our group enables us to assess sweetness exposure within a diet, by profiling foods based on six taste clusters (neutral; salt, umami & fat; sweet and fat; sweet and sour; fat; bitter).

Preference and perceived taste intensity will be assessed during hedonic and sensory evaluation of eight foods; three sweet familiar, three sweet unfamiliar and two salty familiar ones. Foods are solid, semi-solid and liquid. Furthermore, observed food choice and intake during test meals, reported food preferences, reported food cravings, sweet-liker type, glucose homeostasis, body weight, body composition and biomarkers related to diabetes and cardiovascular disease will be assessed. Outcomes will be assessed several times; at baseline (Month 0), during the intervention Month 1, Month 3, Month 6 and in the follow up period (Month 7, Month 10). Compliance will be assessed with 24-hour urine sample and dietary assessment methods (24-hour recalls).

ELIGIBILITY:
Inclusion Criteria:

* Good general health;
* Age 18 - 65 years;
* Body mass index 18.5 - 30 kg/m2;
* Having normal taste ability (assessed with taste strips test);
* Having normal glucose levels in blood (assessed with a finger prick);
* Able to provide informed consent;
* Able to attend Wageningen University, as required for testing.

Exclusion Criteria:

* Diagnosed with diabetes currently or in the past;
* Has been notified to have insulin resistance currently or in the past;
* Diagnosed with endocrine diseases or other metabolic diseases that influence metabolism;
* Diagnosed with eating disorders;
* Diagnosed with taste or smell disorder;
* Pregnant or lactating during the study intervention;
* Gain or loss of more than 3 kg in the last three months prior to study entry;
* Suffering from lack of appetite (self-report);
* Use of medication that may influence study results; such as medication that may affect blood sugar;
* Having a food allergy or/and food intolerance for foods used in the preference testing (e.g. lactose intolerance, celiac disease, egg allergy);
* Consumes more than 14 glasses of alcohol per week;
* Use of soft or hard drugs (e.g. cannabis);
* Student or personnel of Nutrition and Health at Wageningen University;
* Participating in another study/studies or planning to participate in another study.

Specific criteria for withdrawal:

* Pregnancy;
* Weight change of 4 kg or more. In a case of systematic weight change - a subject has gained or lost 4 kg or more at the 3-month period, he/she will be excluded from the study (stop criterion).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Change in preference score. | from month 0 to month 6.
  Measured during preference testing, using Ranking on a scale methodology (scale anchored at 0: Dislike extremely; 50: Neither dislike or like; 100: Like extremely) in a series of test foods.

SECONDARY OUTCOMES:
Change in preference score. | from month 0 to month 1, 3, 7 ad 10.
  Measured during preference testing, using Ranking on a scale methodology (scale anchored at 0: Dislike extremely; 50: Neither dislike or like; 100: Like extremely) in a series of test foods.
Difference in mean liking scores between familiar and unfamiliar foods. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured during preference testing, using Ranking on a scale methodology (scale anchored at 0: Dislike extremely; 50: Neither dislike or like; 100: Like extremely) in a series of test foods.
Change in sensory intensity scores. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured during sensory testing, using 100-unit Visual analogue scale (VAS), (anchored at 0: not sweet/salty at all; 100: Extremely sweet/salty) in a series of test foods.
Change in energy intake. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured during ad-libitum test meal in kcal.
Change in energy intake. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured during ad-libitum test meal in kJ.
Proportion of eaten sweet foods vs. foods from other taste modalities. | Measured at 0, 1, 3, 6, 7 and 10 months
  Measured during ad-libitum test meal in proportions.
Sweet-liker status score. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured on a 100-unit VAS scale (anchored at 0: Dislike; 100: Like).
Food craving questionnaire scores. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured using the Control of eating questionnaire (CoEQ)
Taste preference questionnaire scores. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured using Taste Preference questionnaire (PrefQuest).
Dietary taste patterns. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured with the Taste food frequency questionnaire in frequency.
Dietary taste patterns. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured with the Taste food frequency questionnaire in % of energy coming from each taste cluster.
Dietary taste patterns. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured with the Taste food frequency questionnaire in % of food weight coming from each taste cluster.
Body weight. | Measured at 0, 1, 2, 3, 4, 5, 6, 7 and 10 months.
  Measured with a weighing scale in kg.
Waist-to-hip ratio. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured using a stretch-resistant tape.
% of body fat mass and lean body mass (fat free mass). | Measured at 0, 6 and 10 months.
  Measured with a dual energy x-ray absorptiometry (DEXA).
Variation in interstitial glucose levels. | Measured at 0, 6 and 10 months.
  Measured with glucose monitoring sensor (only measured in a subgroup, of 60 subjects, 20 per intervention arm).
Change in fasting glucose, insulin, total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglycerides levels in blood. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured in blood in mmol/L.
Adverse events. | Measured at 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months.
  Self-reported and monitored.
Concentration of biomarkers in urine related to sugar, low and no calorie sweeteners, protein and salt intake. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured in urine in mg/d.
Intake levels of foods, food groups and macronutrients. | Measured at 0, 1, 2, 3, 4, 5, 6, 7 and 10 months.
  Measured with 24-hour recalls, in kcal/day.
Intake levels of foods, food groups and macronutrients. | Measured at 0, 1, 2, 3, 4, 5, 6, 7 and 10 months.
  Measured with 24-hour recalls, in kJ/day.
Intake levels of foods, food groups and macronutrients. | Measured at 0, 1, 2, 3, 4, 5, 6, 7 and 10 months.
  Measured with 24-hour recalls, in g/day.

OTHER OUTCOMES:
Gender. | Assessed at month 0.
  Self-reported.
Height. | Assessed at month 0.
  Measured with a stadiometer.
Physical activity level. | Measured at 0, 1, 3, 6, 7 and 10 months.
  Measured with the Short Questionnaire to Assess Health enhancing physical activity (SQUASH).
Polymorphisms in the genes related to the sweet taste perception. | Assessed at month 0.
  Genes will be extracted from collected blood samples.
Age. | Assessed at month 0.
  Self-reported.
Medicine usage. | Assessed at month 0.
  Number and type of medicine used, self-reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kees de Graaf, Study Chair — WU; Monica Mars, Principal Investigator — WU
Locations (1):
- Department of Human Nutrition, Wageningen University, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in an article after de-identification will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following the publication. No end date.
Access Criteria: Anyone who wishes to access the data. Individuals who wish to use the data for secondary analysis must contact corresponding authors of respective/specific publications for their approval. They must also reference the source of the data to provide appropriate credit to those who generated it and allow searching for the studies it has supported.

REFERENCES:
- [Background] Cad EM, Tang CS, de Jong HBT, Mars M, Appleton KM, de Graaf K. Study protocol of the sweet tooth study, randomized controlled trial with partial food provision on the effect of low, regular and high dietary sweetness exposure on sweetness preferences in Dutch adults. BMC Public Health. 2023 Jan 11;23(1):77. doi: 10.1186/s12889-022-14946-4. PMID 36627602
- [Derived] Cad EM, Mars M, Pretorius L, van der Kruijssen M, Tang CS, de Jong HB, Balvers M, Appleton KM, de Graaf K. The Sweet Tooth Trial: A Parallel Randomized Controlled Trial Investigating the Effects of A 6-Month Low, Regular, or High Dietary Sweet Taste Exposure on Sweet Taste Liking, and Various Outcomes Related to Food Intake and Weight Status. Am J Clin Nutr. 2026 Jan;123(1):101073. doi: 10.1016/j.ajcnut.2025.09.041. Epub 2025 Nov 27. PMID 41485871

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT04497974/SAP_000.pdf